CLINICAL TRIAL: NCT01806376
Title: A Phase I Study of Subutinib Maleate Capsules on Toleration and Pharmacokinetics
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Collaborators: Fudan University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SBYN-Ⅰ-01
Record Dates: First submitted 2013-03-01; First posted 2013-03-07 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Subutinib Maleate capsules (Experimental): Dose escalation will be dependent on any dose limiting toxicities
  Interventions: Drug: Subutinib Maleate capsules

INTERVENTIONS:
Drug: Subutinib Maleate capsules — Dose escalation will be dependent on any dose limiting toxicities

SUMMARY:
1. purpose: to explore the maximum tolerated dose, dose-limiting toxicity of oral Subutinib Maleate capsules and rational dosage regimen for phase Ⅱ study
2. Experimental Design： A phase Ⅰ study of single-center
3. Test drug: Subutinib Maleate capsules
4. Sample size≥20

DETAILED DESCRIPTION:
The primary objective of this study is to explore the maximum tolerated dose, dose-limiting toxicity of oral Subutinib Maleate capsules and rational dosage regimen for phase Ⅱ study, to investigate the pharmacokinetics of single and multiple oral doses of Subutinib Maleate capsules.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have histologically or cytologically confirmed solid tumors
* Subjects who have failed standard effective therapy or have a diagnosis for which no standard effective treatment is available;
* Aged 18 to 70 years old; Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2; Life expectancy greater than 3 months;
* If the subject has been given other chemotherapy drugs, it's necessary to discontinue them more than 4 weeks. If the chemotherapy drugs are Nitrosoureas and Mitomycin C, it's necessary to discontinue them more than 6 weeks. If the subject has accepted major surgery, it's necessary to wait more than 4 weeks before the subject participating in this study.
* Blood test: Hb≥100g/L(no blood transfusion within 14 days); ANC≥1.5×109/L, PLT≥100×109/L
* Biochemistry: TBIL and ALT and AST and Cr are in normal range, or creatinine clearance ≥60ml/min; Triglyceride≤3.0mmol/L; Cholesterol ≤7.75mmol/L.
* Doppler ultrasound measurement: LVEF ≥ LLN
* Female subjects should agree to take contraceptives during the study and within 6 months after the study (such as intrauterine device [IUD], contraceptive drugs or condoms); within 7 days before they enter the study, their serum or human chorionic gonadotropin should be negative, and must be in the non-lactation period; male subjects should agree to take contraceptives during the study and within 6 months after the study.
* The subject is willing to participate in this study, and he/she has signed the Informed Consent Form, with good compliance.

Exclusion Criteria:

* The subject has participated in other drug clinical research in the past 4 weeks.
* The subject is accompanied with several factors which will influence the investigational drug administration orally, such as inability to swallow or after gastrointestinal resection or chronic diarrhea or intestinal obstruction.
* Central nervous system metastasis definitely.
* The subject is suffering from hypertension or myocardial ischemia or myocardial infarction or arrhythmia (including QT interval≥440ms) or Grade I heart failure.
* If the subject's systolic BP is over 140mmhg, with diastolic BP over 90mmhg, or the subject's blood pressure is well-controlled, he/she is not permitted to enroll in this study as well.
* The subject's urinalysis displays that urinary protein ≥ ++ , combined with 24-hour urinary protein > 1.0g.
* The subject's is suffering from wounds or fractures which can not be cured for long time.
* Abnormal coagulation: The subject has bleeding tendency such as active peptic ulcer or the subject is receiving thrombolytic or anticoagulant therapy.
* There are pre-dosing arterial/venous thrombotic events on this subject, such as cerebrovascular accident (including TIA) or deep vein thrombosis or pulmonary embolism.
* The subject is accepting anticoagulants or vitamin K antagonists such as warfarin or heparin or analogue therapy; If the subject's INR ≤ 1.5, he/she is allowed to use small doses of warfarin (1mg oral q d) or small doses of aspirin(less than 100mg each day), and the purpose of the treatment should be prevention.
* Abnormal thyroid function.
* There is history of mental drug abuse occurred in the subject, or the subject is suffering from mental disorders.
* There is history of immunodeficiency occurred in the subject, including HIV positive or other acquired or congenital immunodeficiency diseases, or the subject has accepted organ transplant before.
* Lung squamous cell carcinoma.
* The subject has received small molecule targeted drug therapy of inhibition of VEGFR-2 and PDGFRβ
* According to the investigator's judgment, there are concomitant diseases which will seriously do harm to the subject's safety or obstruct the subject to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity， maximum tolerated dose. | 2 months

SECONDARY OUTCOMES:
Pharmacokinetics | 2 months
  Subutinib Maleate pharmacokinetic parameters , include AUC, Cmax, Tmax, and t1/2
Pharmacodynamics | 2 months
  The response of Subutinib Maleate on tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Li jin, doctor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China